CLINICAL TRIAL: NCT04239170
Title: An Open-lable, Single Arm, Phase 2 Study of Camrelizumab(SHR-1210) Combined With GEMOX in Patients With Relapsed or Refractory Hodgkin Lymphoma Who Will Receive ASCT
Brief Title: Camrelizumab(SHR-1210) Combined With GEMOX in Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Party secretary of Cancer Hospital of Peking University, Director of Internal Medicine, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-GEMOX-IIT-HL
Record Dates: First submitted 2020-01-20; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — camrelizumab; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab(SHR-1210) Combined With GEMOX (Experimental)
  Interventions: Drug: Camrelizumab(SHR-1210)

INTERVENTIONS:
Drug: Camrelizumab(SHR-1210) — Camrelizumab(SHR-1210): A humanized monoclonal immunoglobulin
  Other Names: GEMOX(Gemcitabine, Oxaliplatin)

SUMMARY:
This is an open-label, single arm, Phase 2 study to evaluate efficacy and safety of PD1 inhibitor Camrelizumab(SHR-1210) combined with Gemox in patients with relapsed and refractory hodgkin lymphoma who will receive ASCT.Efficacy will be assessed according to 2014 Lugano criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed classic Hodgkin's lymphoma ;
2. Relapsed or refractory cHL and meet any of the following criterions:a)did not achieve remission or progression and will receive autologous hematopoietic stem cell transplantation.b)receive no more than 3 lines of systemic chemotherapy.
3. Subjects enrolled have measurable lesion(s) according to Lugano 2014 criteria
4. ECOG performance status of 0 or 1;
5. Life expectancy ≥ 12 weeks.;
6. Adequate laboratory parameters during the screening period as evidenced by the following:

   1. Hemoglobin ≥ 90 g/L;
   2. Absolute neutrophil count ≥ 1.5 × 109/L ;
   3. Platelets ≥ 100 × 109/L;
   4. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN),
   5. ALT and AST ≤ 2.5×ULN
   6. Serum Creatinine ≤1.25×ULN or Creatinine clearance≥60 mL/min;
   7. Coagulation function index：INR ≤1.5×ULN，APTT≤1.5×ULN
7. Women of childbearing potential（WOCBP）with pregnancy test negative within 7 days before entering the group and consent to employ a highly effective method of birth control/contraception to prevent pregnancy for at least 1 year after receiving the last dose of study treatment; Male subjects with WOCBP partner should receive Surgical sterilization or consent to employ a highly effective method of birth control/contraception to prevent pregnancy for at least 1 year after receiving the last dose of study treatment.
8. Able to understand and sign an informed consent form (ICF).

Exclusion Criteria:

1. Known nodular lymphoma predominant Hodgkin lymphoma
2. History and complication as follows,

   1. Active, known or suspected autoimmune disease. Subjects who were in a stable state without systemic immunosuppressive therapy were admitted
   2. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic corticosteroids > 10 mg/day topical prednisone or equivalent are prohibited within 2 weeks before entering the group
   3. Received anti-tumor vaccines or other anti-tumor therapy with immune stimulation within 3 months before the first dose of trial drugs.
   4. Prior exposure to any PD-1/PD-L1/PD -L 2 or CTLA -4 antibody . Or prior exposure to GEMOX but PD.
   5. Participating in other clinical studies or less than 4 weeks before the end of a clinical trial.
   6. Known and highly Suspicion of interstitial pneumonia.
   7. Other active malignancies that required treating. (subjects with skin basal cell carcinoma, superficial bladder cancer, skin squamous cell carcinoma or cervical carcinoma who had no disease recurrence within 5 years after the start of treatment were excluded).
   8. Received chemotherapy, radiotherapy,immunotherapy, including topical therapy within 4 weeks. Previous anti-tumor therapy related adverse reactions (except hair loss) did not recover to CTCAE ≤1.
   9. Prior allo-HSCT.
   10. Impact of major surgery or severe trauma had been eliminated for less than 28 days
   11. Active pulmonary tuberculosis.
   12. Severe acute or chronic infection requiring systemic therapy.
   13. Suffering from high blood pressure, and cannot be well controlled by antihypertensive drugs (systolic pressure ≥ 140 mmHg or diastolic pressure ≥ 90 mmHg)
   14. Suffering from heart failure (New York Heart Association standard III or IV). Uncontrolled coronary artery disease and arrhythmia although given appropriate medical treatment. History of myocardial infarction within 6 months.
   15. Three months before randomization, there were significant bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer, stool occult blood test is ++ at baseline and above, or vasculitis
3. Laboratory test

   1. Known HIV positive or known AIDS.
   2. Untreated active hepatitis: Hepatitis B(HBsAg positive and HBV DNA≥500IU/mL), and hepatitis C(HCV RNA positive, abnormal liver function) ,Hepatitis B and hepatitis C infection in common.
4. Other factors that may lead to the study termination, such as severe disease or abnormal laboratory tests or family or social factors affecting subjects safety or test data and sample collection.
5. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Complete Response | From first patient first visit to 3 month after last patient first visit
  Based on Lugano 2014 criteria

SECONDARY OUTCOMES:
Objective Response Rate | From first patient first visit to 3 month after last patient first visit
  Rate of subjects achieved complete response plus partial response in all evaluable subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Ping L, Song Y, Tang Y, Zheng W, Liu W, Ying Z, Zhang C, Wu M, Feng F, Lin N, Tu M, Zhu J, Xie Y. Camrelizumab plus gemcitabine and oxaliplatin for relapsed or refractory classical Hodgkin lymphoma: a phase II trial. BMC Med. 2024 Mar 7;22(1):107. doi: 10.1186/s12916-024-03329-8. PMID 38454451